CLINICAL TRIAL: NCT04697628
Title: A Randomized, Open-Label, Phase 3 Trial of Tisotumab Vedotin vs Investigator's Choice Chemotherapy in Second- or Third-Line Recurrent or Metastatic Cervical Cancer
Brief Title: Tisotumab Vedotin vs Chemotherapy in Recurrent or Metastatic Cervical Cancer
Acronym: innovaTV 301
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNTV-003; C5721002 (Other: Alias Study Number); 2023-503813-31-01 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: Seattle Genetics
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tisotumab vedotin; Topotecan; Vinorelbine; Gemcitabine; Irinotecan; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tisotumab vedotin (Experimental): Tisotumab vedotin monotherapy
  Interventions: Drug: tisotumab vedotin
- Chemotherapy (Active Comparator): Investigator's choice of one chemotherapy treatment (topotecan, vinorelbine, gemcitabine, irinotecan, or pemetrexed)
  Interventions: Drug: topotecan; Drug: vinorelbine; Drug: gemcitabine; Drug: irinotecan; Drug: pemetrexed

INTERVENTIONS:
Drug: tisotumab vedotin — 2.0 mg/kg every 3 weeks (Q3W)
  Other Names: TIVDAK; PF-08046057
  Arms: Tisotumab vedotin
Drug: topotecan — 1 or 1.25 mg/m2 intravenous (IV) on Days 1 to 5, every 21 days
  Arms: Chemotherapy
Drug: vinorelbine — 30 mg/m2 IV on Days 1 and 8, every 21 days
  Arms: Chemotherapy
Drug: gemcitabine — 1000 mg/m2 IV on Days 1 and 8, every 21 days
  Arms: Chemotherapy
Drug: irinotecan — 100 or 125 mg/m2 IV weekly for 28 days, every 42 days
  Arms: Chemotherapy
Drug: pemetrexed — 500 mg/m2 IV on Day 1, every 21 days
  Arms: Chemotherapy

SUMMARY:
This trial is being done to find out whether tisotumab vedotin works better than chemotherapy to treat cervical cancer. People in this study have cervical cancer that has spread to other parts of the body (metastatic) or has come back after being treated (recurrent).

Participants in this trial will be randomly assigned to one of two groups. One group will be treated with tisotumab vedotin. Participants in the other group will get one of five different chemotherapy drugs (topotecan, vinorelbine, gemcitabine, pemetrexed, or irinotecan). Participants and their doctors will know which group they are in. Participants in the chemotherapy group will decide with their study doctor which drug they will take.

ELIGIBILITY:
Inclusion Criteria

* Has recurrent or metastatic cervical cancer with squamous cell, adenocarcinoma, or adenosquamous histology, and:
* Has experienced disease progression during or after treatment with a standard of care systemic chemotherapy doublet, or platinum-based therapy (if eligible), defined as either:

  * paclitaxel + cisplatin + bevacizumab + anti-PD-(L)1 agent, or
  * paclitaxel + carboplatin + bevacizumab + anti-PD-(L)1 agent, or
  * paclitaxel + topotecan/nogitecan + bevacizumab + anti-PD-(L)1 agent
* Note: In cases where bevacizumab and/or anti-PD-(L)1 agent is not a standard of care therapy or the participant was ineligible for such treatment according to local standards, prior treatment with bevacizumab and/or anti-PD-(L)1 agent is not required.
* Has received 1 or 2 prior systemic therapy regimens for recurrent and/or metastatic cervical cancer. Chemotherapy administered in the adjuvant or neoadjuvant setting, or in combination with radiation therapy, should not be counted as a systemic therapy regimen. Single agent therapy with an anti-PD(L)1 agent for r/mCC cancer should be counted.
* Measurable disease according to RECIST v1.1 as assessed by the investigator.
* Has ECOG performance status of 0 or 1 prior to randomization.
* Has life expectancy of at least 3 months.

Exclusion Criteria

* Has primary neuroendocrine, lymphoid, sarcomatoid, or other histologies not mentioned as part of the inclusion criteria above.
* Has clinically significant bleeding issues or risks. This includes known past or current coagulation defects leading to an increased risk of bleeding; diffuse alveolar hemorrhage from vasculitis; known bleeding diathesis; ongoing major bleeding; trauma with increased risk of life-threatening bleeding or history of severe head trauma or intracranial surgery within 8 weeks of trial entry.
* Has any history of intracerebral arteriovenous malformation, cerebral aneurysm, or stroke (transient ischemic attack >1 month prior to screening is allowed).
* Active ocular surface disease or a history of cicatricial conjunctivitis or inflammatory conditions that predispose to cicatrizing conjunctivitis (e.g. Wagner syndrome, atopic keratoconjunctivitis, autoimmune disease affecting the eyes), ocular Stevens-Johnson syndrome or toxic epidermal necrolysis, mucus pemphigoid, and participants with penetrating ocular transplants. Cataracts alone is not an exclusion criterion.
* Major surgery within 4 weeks or minor surgery within 7 days prior to the first study treatment administration.
* Peripheral neuropathy ≥grade 2.
* Any prior treatment with monomethyl auristatin E (MMAE)-containing drugs.

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 502 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2026-05-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (209):
- United States (52):
  - Arizona Oncology Associates, PC - HAL, Glendale, Arizona
  - Arizona Oncology Associates P.C. - NAHOA, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - University of California Irvine Health, Irvine, California
  - UC Irvine Health (Investigator Site File Location), Orange, California
  - University of California Irvine Health, Orange, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Attn. Becky Champion, PharmD, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Norton Women's & Children's Hospital, Louisville, Kentucky
  - Willis-Knighton Cancer Center Infusion Center, Shreveport, Louisiana
  - Willis-Knighton Physician Network/ Hematology-Oncology Associates, Shreveport, Louisiana
  - Willis-Knighton Physician Network/WK Gynecologic Oncology Associates, Shreveport, Louisiana
  - Minnesota Oncology Hematology PA, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A, Edina, Minnesota
  - Minnesota Oncology Hematology, P.A, Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A, Minneapolis, Minnesota
  - Minnesota Oncology Hematology, P.A, Saint Paul, Minnesota
  - St. Dominic- Jackson Memorial Hospital Pharmacy Attn: Richard Wakefield, Jackson, Mississippi
  - Washington University School of Medicine- Obstetrics & Gynecology [Academic Offices], St Louis, Missouri
  - Washington University School of Medicine [Patient Clinics], St Louis, Missouri
  - Washington University School of Medicine-Obstetrics & Gynecology, St Louis, Missouri
  - NewYork Presbyterian - Brooklyn Methodist Hospital, Brooklyn, New York
  - NewYork Presbyterian - Queens, Flushing, New York
  - NewYork Presbyterian - Queens, Forest Hills, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone., New York, New York
  - NYU Langone Medical Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic Fail·view Hospital, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital- Moll Cancer Center lnvestigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic., Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, OSU Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - VCU Health, Investigational Drug Service (ATTN: Henly Deutsch, RPh), Richmond, Virginia
- Argentina (4):
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires, Buenos Aires F.D.
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Fundacion CENIT para la lnvestigacion en Neurociencias, Buenos Aires
  - IONC - Instituto Oncologico de Cordoba, Córdoba
- Radiologie - Diagnosezentrum Urania, Vienna, Austria
- Belgium (7):
  - Cliniques Universitaires Saint Luc, Brussels, Brabant
  - Institut Jules Bordet, Anderlecht
  - ZNA Middelheim, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven-Campus Gasthuisberg, Leuven
  - CHU de Liege - Sart Tilman, Liège
  - CHU UCL Namur-Site St-Elisabeth, Namur
- Brazil (9):
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ljui, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital de Sao Lucas da Pontificia Universidade CatoIica do Rio Grande do Sul -PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - A Beneficencia Portuguesa de Sao Paulo - BP Mirante, São Paulo, São Paulo
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba/PR
  - lnstituto Nacional de Cancer Jose Alencar Gomes da Silva - INCA- Coordenacao de Pesquisa Clinica, Rio de Janeiro
  - CIPE Centro Internacional de Pesquisa - AC Camargo Cancer Center - CAPEC Centro de Apoio a Pesquisa, São Paulo
  - lnstituto Brasileiro de Controle do Cancer - IBCC, São Paulo
- Canada (6):
  - Cross Cancer Institute Cancer Committee, Edmonton, Alberta
  - BC Cancer - Vancouver Center, Vancouver, British Columbia
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- China (27):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital., Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College,Huazhong University of science and Technology, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital., Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital., Xi'an, Shaanxi
  - Affiliated Cancer Hospital of Shandong First Medical University (Shandong Cancer Hospital&Institute), Jinan, Shandong
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Cancer Hospital Chinese Academy of Medical Sciences (CAMS), Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Obstetrics And Gynecology Hospital, Capital Medical University Bejing Maternal and Child, Beijng
  - The Second Hospital of Dalian Medical University, Dalian
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning
  - Shanghai General Hospital, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
- Czechia (4):
  - Onkologická ambulance Gynekologicko-porodnická klinika FN Brno, Brno
  - Onkologicka klinika FN Olomouc, Olomouc
  - Gynekologicko-porodnicka klinika 1. lekarske fakulty a Vseobecne fakultni nemocnice, Prague
  - Fakultni nemocnice Bulovka, Gynekologicko-porodnicka klinika, Praha 8-Liben
- Turku University Hospital, Lighthouse Hospital, Gynecology Outpatient Clinic, Turku, Finland
- France (9):
  - Centre Hospitalier Regional et Universitaire de Besancon - Hopital Jean-Minjoz, Besançon
  - lnstitut Bergonie Centre Regional de Lutte contre le Cancer, Bordeaux
  - HPC -Service d'Oncologie Medicale, Nantes
  - HPC -Service Pharmacie, Nantes
  - Groupe Hospitalier Diaconesses Croix-Saint-Simon, Paris
  - Hopital Prive des Cotes d'Armor - Centre CARIO, Plérin
  - Institut de Cancerologie de Strasbourg, Strasbourg
  - lnstitut Claudius Regaud - IUCT-O, Toulouse
  - lnstitut Gustave Roussy, Villejuif
- Germany (8):
  - Universitaetsklinikum Hamburg-Eppendorf (UKE), Hamburg, North Rhine-Westphalia
  - KEM / Evang. Kliniken Essen-Mitte gGmbH, Essen
  - University Hospital Essen, Clinic for Obstetrics and Gynecology, Essen
  - KEM / Evang. Kliniken Essen-Mitte gGmbH Evang. Krankenhaus Essen Warden, Essen
  - UKE, Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Augenklinik der LMU, München
  - LMU Klinikum Klinik und Poliklinik fur Frauenheilkunde und Geburtshilfe, München
  - LMU Klinikum, München
- Hungary (6):
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét, Bács-Kiskun county
  - National Institute of Oncology,Department of Gynecology, Budapest, Other
  - Debreceni Egyetem Klinikai Kozpont, Szuleszeti es Nogyogyaszati Klinika, Debrecen
  - Debreceni Egyetem, Klinikai Kozpont, Orvosi Kepalkoto Klinika-Radiologia, Debrecen
  - Debreceni Egyetem, Klinikai Kozpont, Szemklinika, Debrecen
  - Scanomed Kft., Debrecen
- Italy (4):
  - Servizio di Farmacia, Milan, Milan
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome, Other
  - Oncologia di Vicenza - Ospedale San Bortolo, Vicenza, Veneto
  - Unita Farmaci Antiblastici, Vicenza, Veneto
- Japan (26):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Jikei University Kashiwa Hospital, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Ota-Shi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Nippon Medical School Musashikosugi Hospital, Kawasaki, Kanagawa
  - University of the Ryukyus Hospital, Ginowan, Okinawa
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima City Hospital, Kagoshima
  - Yokohama City University Hospital, Kanagawa
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - The Cancer Institute Hospital of JFCR, Tokyo
- Oncologico Potosino, San Luis Potosí City, Mexico
- Netherlands (7):
  - Erasmus Medisch Centrum Daniel Den Hoed, Rotterdam, South Holland
  - Amsterdam UMC, Department of Oncology, Amsterdam
  - MUMC+ Medical Oncology, Maastricht
  - Radboud UMC, afd Medische Oncologie (hp452), Nijmegen
  - Erasmus MC Clinical Trial Center, Rotterdam
  - Erasmus MC Interne Oncologie, Rotterdam
  - UMC Utrecht - Trialbureau Medische Oncologie, Utrecht
- Norway (2):
  - Oslo Universitetssykehus HF, Radiumhospitalet, Oslo
  - Sykehusapoteket Oslo, Radiumhospitalet, Oslo
- RCI 621 Hospital Maria Auxiliadora Unidad de investigacion en Oncologia, Lima, Peru
- Białostockie Centrum Onkologii, Bialystok, Poland
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (11):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si, Chungcheongnam-do
  - Soon Chun Hyang University Hospital Cheonan, Cheonan-si, Chungcheongnam-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Cneter, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Changwon Hospital, Changwon-si, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Clínica Universidad de Navarra - Pamplona, Pamplona, Navarra, Comunidad Foral de
  - Clinica Universitaria de Navarra (sede Navarra), Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Universitaria de Navarra (sede Madrid), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Clinico Valencia, INCLIVA, Valencia
- Sweden (3):
  - Kliniska forskningsenheten, VE Onkologi och Stralningsfysik, Lund
  - Skanes University Hospital, Lund
  - ApoEx AB, Kliniska provningar, Malmo
- Taiwan (4):
  - Clinical Pharmacy, Mackay Memorial Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan City Singapore
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge, England
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vergote I, Gonzalez-Martin A, Fujiwara K, Kalbacher E, Bagameri A, Ghamande S, Lee JY, Banerjee S, Maluf FC, Lorusso D, Yonemori K, Van Nieuwenhuysen E, Manso L, Woelber L, Westermann A, Covens A, Hasegawa K, Kim BG, Raimondo M, Bjurberg M, Cruz FM, Angelergues A, Cibula D, Barraclough L, Oaknin A, Gennigens C, Nicacio L, Teng MSL, Whalley E, Soumaoro I, Slomovitz BM; innovaTV 301/ENGOT-cx12/GOG-3057 Collaborators. Tisotumab Vedotin as Second- or Third-Line Therapy for Recurrent Cervical Cancer. N Engl J Med. 2024 Jul 4;391(1):44-55. doi: 10.1056/NEJMoa2313811. PMID 38959480
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTV-003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with recurrent/metastatic cervical cancer (rCC/mCC) who received 1 or 2 prior lines of systemic therapy for their recurrent or metastatic disease were included.
Pre-assignment Details: A total of 660 participants were screened of which 158 participants failed screening and 502 participants were enrolled in the study.
Groups:
- Tisotumab Vedotin: Participants with rCC/mCC were administered tisotumab vedotin 2.0 milligram per kilogram (mg/kg) as an intravenous (IV) infusion once every 3 weeks (Q3W).
- Chemotherapy: Participants with rCC/mCC were treated with investigator's choice of chemotherapy which included either topotecan 1 or 1.25 milligram per meter square [mg/m^2] IV on Days 1 to 5, every 21 days or vinorelbine 30 mg/m^2 IV on Days 1 and 8, every 21 days or gemcitabine 1000 mg/m^2 IV on Days 1 and 8, every 21 days or irinotecan 100 or 125 mg/m^2 IV weekly for 28 days, every 42 days or pemetrexed 500 mg/m^2 on Day 1, every 21 days.
Period: Overall Study
Arm/Group | Tisotumab Vedotin | Chemotherapy
Started | 253 | 249
Treated | 250 | 239
Completed | 114 (Completers include participants who died from any cause.) | 131 (Completers include participants who died from any cause.)
Not Completed | 139 | 118
Not completed — Withdrawal by Subject | 17 | 23
Not completed — Lost to Follow-up | 0 | 4
Not completed — On-going in study | 122 | 91

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants. Participants were included in the treatment group assigned at randomization regardless of any actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tisotumab Vedotin | Chemotherapy | Total
Number analyzed (Participants) | 253 | 249 | 502
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (11.8) | 51.0 (11.6) | 51.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 249 | 502
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race is reported.
  Participants
    Race: White | 122 | 122 | 244
    Race: Asian | 90 | 90 | 180
    Race: American Indian or Alaska Native | 7 | 7 | 14
    Race: Black or African American | 4 | 6 | 10
    Race: Other | 2 | 1 | 3
    Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Race: Not Reported | 19 | 17 | 36
    Race: Unknown | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity is reported.
  Participants
    Ethinicity: Not of Hispanic or Latino/a, or Spanish Origin | 176 | 177 | 353
    Ethinicity: Hispanic or Latino/a, or of Spanish Origin | 52 | 50 | 102
    Ethinicity: Not Reported | 19 | 17 | 36
    Ethinicity: Unknown | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive.
Time Frame: From randomization to date of death due to any cause or censoring date, whichever occurred first (maximum up to 25 months)
Population: ITT analysis set included all randomized participants. Participants were included in the treatment group assigned at randomization regardless of any actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 253 | 249
Months | 11.5 [9.8 to 14.9] | 9.5 [7.9 to 10.7]
Statistical Analysis 1: Comparison: Tisotumab Vedotin vs Chemotherapy; Test type: Superiority; p = 0.0038, Stratified log-rank test — Two-sided p-value calculated from stratified log-rank test; Cox Proportional Hazard = 0.70, 95% CI 2-sided [0.54 to 0.89] — Hazard Ratio (HR) was calculated from Cox proportional hazards model and Efron method was used in handling ties and computed using stratification factors at randomization

2. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigator
Description: PFS per investigator was defined as the time from the date of randomization to the first documentation of disease progression (PD) as assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, or death due to any cause, whichever occurred earlier. PD: at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). Participants without evidence of radiographic disease progression or death were censored at the date of last adequate tumor assessment prior to data cut-off date or start of new anti-cancer therapy. Participants with disease progression or death that occurred after 2 or more missed scans were censored at the last adequate tumor assessment prior to missed scans. Participants without post-baseline scan data were censored at the day of randomization.
Time Frame: From the date of randomization to first documentation of PD or death due to any cause, or censoring date whichever occurred first (maximum up to 25 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 253 | 249
Months | 4.2 [4.0 to 4.4] | 2.9 [2.6 to 3.1]
Statistical Analysis 1: Comparison: Tisotumab Vedotin vs Chemotherapy; Test type: Superiority; p < 0.0001, Stratified log-rank test — Two-sided p-value calculated from stratified log-rank test; Cox Proportional Hazard = 0.67, 95% CI 2-sided [0.54 to 0.82] — HR was calculated from Cox proportional hazards model and Efron method was used in handling ties and computed using stratification factors at randomization

3. Secondary Outcome: Confirmed Objective Response Rate (ORR) as Assessed by Investigator
Description: Confirmed objective response rate was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v.1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The minimum criteria for stable disease (SD) duration are defined as ≥ 5 weeks after the date of randomization. For a response to be considered as confirmed, the subsequent response had to be at least 4 weeks after the initial response. Two-sided 95% exact confidence interval (CI) was computed using the Clopper-Pearson method.
Time Frame: From the date of randomization until date of confirmed CR or PR (maximum up to 25 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 253 | 249
Percentage of participants | 17.8 [13.3 to 23.1] | 5.2 [2.8 to 8.8]
Statistical Analysis 1: Comparison: Tisotumab Vedotin vs Chemotherapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.0, 95% CI 2-sided [2.1 to 7.6] — OR calculated using Cochran-Mantel-Haenszel (CMH) method controlling for stratification factors at randomization

4. Secondary Outcome: Time-to-Response (TTR) as Assessed by the Investigator
Description: TTR was defined as the time from the randomization date to the date of the first confirmed objective response (CR or PR that was subsequently confirmed). CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to date of date of the first confirmed objective response (maximum up to 25 months)
Population: ITT analysis set included all randomized participants. Participants were included in the treatment group assigned at randomization regardless of any actual treatment received. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Only participants who achieved a confirmed CR or PR based on investigator assessment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 45 | 13
Months | 1.58 [1.2 to 4.5] | 1.74 [1.2 to 3.9]

5. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment
Description: DOR was defined as the time from the date of the first confirmed objective response (CR or PR that was subsequently confirmed) to the date of the first documented PD per RECIST v1.1 or death from any cause, whichever occurred first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of first documented response of CR or PR to the first documented PD or death from any cause, whichever occurred first (maximum up to 25 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 45 | 13
Months | 5.3 [4.2 to 8.3] | 5.7 [2.8 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with event.

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment and with onset date on or before 30 days after the last dose of study treatment.
Time Frame: From start of treatment up to 30 days after last dose of study treatment (up to 25 months)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment (tisotumab vedotin or chemotherapy).
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin | Chemotherapy
Number analyzed (Participants) | 250 | 239
Participants | 246 | 237

7. Secondary Outcome: EuroQOL Five Dimensions Five Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L questionnaire is a 5-item self-reported measure of functioning and well-being, which assesses 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems). Responses to the 5 items are then converted to a weighted health state index (utility score) based on values derived from general population samples. This health utility score is between 0 and 1, where 0 is death and 1 is perfect health.
Time Frame: From start of treatment until end of follow-up
Reporting Status: Not Posted, anticipated posting 2027-02

8. Secondary Outcome: EQ-5D Visual Analog Scale (VAS) Scores
Description: EQ5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state) ; higher scores indicate a better health state.
Time Frame: From start of treatment until end of follow-up
Reporting Status: Not Posted, anticipated posting 2027-02

9. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Total Score
Description: The EORTC-QLQ-C30 questionnaire is composed of 30 questions for which the answers ranges either from 1 (not at all) to 4 (very much) for items 1 to 28, or from 1 (very poor) to 7 (excellent) for items 29 to 30. The EORTC QLQ-C30 scale scores will be calculated using the EORTC QLQ-C30 Scoring Manual. These include 5 functional scales, 3 symptom scales, a global health status/QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items (i.e., no item occurs in more than one scale). All of the scales and single-item measures range in score from 0 to 100, with a high scale score representing a higher response level (e.g., a high level of functioning, a high QoL, or a high level of symptomatology/problems)
Time Frame: From start of treatment until end of follow-up
Reporting Status: Not Posted, anticipated posting 2027-02

10. Secondary Outcome: EORTC Quality of Life Questionnaire Cervical Cancer Module (QLQ-CX24) Total Scores
Description: The EORTC QLQ-CX24 questionnaire is meant for use among cervical cancer participants varying in disease stage and treatment modality. The EORTC-QLQ-CX24 questionnaire is composed of 24 questions for which the answers ranged from 1 (Not at all) to 4 (Very much). Four functional scales and 5 symptom scales will be calculated using the EORTC QLQ-CX24 Scoring Manual. The 9 scores computed from the EORTC-QLQ-CX24 questionnaire will be summarized by treatment arm using descriptive statistics.
Time Frame: From start of treatment until end of follow-up
Reporting Status: Not Posted, anticipated posting 2027-02

ADVERSE EVENTS:
Time Frame: For All-Cause Mortality: From randomization to date of death due to any cause (up to 25 months); For SAEs and non-SAEs: From start of treatment up to 30 days after last dose of study treatment (approximately up to 25 months)
Description: Same event may appear as both other (non-serious adverse event [non-SAE]) and SAE; however, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Data for all-cause mortality was collected for ITT analysis set, data for SAE and non-SAE were collected for safety analysis set.
Arm/Group | Tisotumab Vedotin | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 123/253 | 140/249
Serious Adverse Events (participants affected / at risk) | 82/250 | 94/239
Other Adverse Events (participants affected / at risk) | 233/250 | 223/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisotumab Vedotin (N=250) | Chemotherapy (N=239)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 10 (12)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 8 (10)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (7) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Truncus coeliacus thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 3 (3) | 4 (4)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 3 (4)
Pyelonephritis acute (Infections and infestations) | 2 (3) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (12) | 17 (21)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 5 (5)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 7 (7)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (5) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisotumab Vedotin (N=250) | Chemotherapy (N=239)
Anaemia (Blood and lymphatic system disorders) | 56 (69) | 119 (160)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 16 (24)
Neutropenia (Blood and lymphatic system disorders) | 15 (18) | 52 (119)
Dry eye (Eye disorders) | 33 (41) | 1 (1)
Keratitis (Eye disorders) | 39 (53) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 30 (36) | 21 (25)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 12 (15)
Constipation (Gastrointestinal disorders) | 59 (68) | 39 (40)
Diarrhoea (Gastrointestinal disorders) | 53 (72) | 36 (45)
Nausea (Gastrointestinal disorders) | 83 (101) | 93 (140)
Vomiting (Gastrointestinal disorders) | 42 (56) | 43 (61)
Asthenia (General disorders) | 40 (49) | 38 (52)
Fatigue (General disorders) | 29 (37) | 36 (41)
Oedema peripheral (General disorders) | 9 (9) | 29 (30)
Pyrexia (General disorders) | 40 (54) | 47 (76)
COVID-19 (Infections and infestations) | 13 (13) | 9 (9)
Conjunctivitis (Infections and infestations) | 77 (106) | 1 (1)
Urinary tract infection (Infections and infestations) | 26 (35) | 25 (36)
Alanine aminotransferase increased (Investigations) | 17 (23) | 26 (31)
Aspartate aminotransferase increased (Investigations) | 16 (18) | 27 (34)
Neutrophil count decreased (Investigations) | 3 (4) | 21 (37)
Platelet count decreased (Investigations) | 0 (0) | 13 (19)
Weight decreased (Investigations) | 24 (26) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 59 (68) | 41 (50)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (17) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (20) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19) | 20 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 8 (8)
Headache (Nervous system disorders) | 11 (11) | 13 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 70 (75) | 6 (7)
Insomnia (Psychiatric disorders) | 19 (21) | 12 (12)
Haematuria (Renal and urinary disorders) | 17 (22) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 6 (6) | 12 (12)
Vaginal haemorrhage (Reproductive system and breast disorders) | 21 (21) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 21 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 14 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 65 (79) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 61 (64) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (39) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT04697628/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT04697628/SAP_001.pdf